CLINICAL TRIAL: NCT04088292
Title: Low Dose Thrombolysis, Ultrasound Assisted Thrombolysis or Heparin for Intermediate High Risk Pulmonary Embolism
Acronym: STRATIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev and Gentofte Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Hillerod Hospital, Denmark (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Jesper Kjaergaard, Sponsor, Primary investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STRATIFY-1
Record Dates: First submitted 2019-09-09; First posted 2019-09-12 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator; Powders; Solutions

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 1:1:1 allocation to treatment strata
Who Masked: Outcomes Assessor
Masking Description: Primary endpoint will be assessed by assessor blinded to the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- USAT + low dose thrombolysis (Active Comparator): UltraSound Assisted Thrombolysis (USAT) with low dose thrombolysis (20 mg of rtPA, Alteplase) over 6 hours plus unfractionated heparin (UFH) or low molecular weight heparin (LMWH) within 12 hours of randomization
  Interventions: Drug: Alteplase 20 Mg Powder for Solution for Injection Vial; Device: Ultrasound assisted Thrombolysis
- Low dose thrombolysis (Active Comparator): Intravenous low dose thrombolysis (20 mg of rtPA, Alteplase) over 6 hours plus UFH or low molecular weight heparin (LMWH).
  Interventions: Drug: Alteplase 20 Mg Powder for Solution for Injection Vial
- Heparin alone (No Intervention): UFH or low molecular weight heparin (LMWH) only (with option for conventional thrombolysis according to local protocols for hemodynamic deterioration)

INTERVENTIONS:
Drug: Alteplase 20 Mg Powder for Solution for Injection Vial — Low dose alteplase delivered IV or bu Ultrasound Assisted Thrombolysis device
  Arms: Low dose thrombolysis; USAT + low dose thrombolysis
Device: Ultrasound assisted Thrombolysis — Ultrasound assisted thrombolysis (USAT)
  Arms: USAT + low dose thrombolysis

SUMMARY:
Open label clinical randomized trial comparing three strategies for managing acute intermediate-high risk pulmonary embolism

DETAILED DESCRIPTION:
Trial acronym: STRATIFY Background: Intermediate-high risk pulmonary embolism (PE) is associated with a significant risk of death or hemodynamic deterioration. The optimal treatment strategy should balance efficacy in reducing thrombus burden and hemodynamic compromise with risk of complications, in particular bleeding. Previous studies have investigated conventional high-dose, short term thrombolysis by (rtPA), finding a reduction in risk hemodynamic deterioration, but no reduction in mortality and a substantial increase in significant bleeding complications.

Catheter based techniques and low dose thrombolysis may offer lower risk of complication with reasonable efficacy. Such studies have not been performed in RCTs with a reasonable sample size, and no study have compared low dose intravenous thrombolysis and catheter based techniques.

The current trial addresses this paucity of data by randomizing patients to one of three treatment modalities:

Intervention: 1:1:1 randomization, stratified for site to

* UltraSound Assisted Thrombolysis (USAT) with low dose thrombolysis (20 mg of rtPA, Alteplase) over 6 hours plus unfractionated heparin (UFH) or low molecular weight heparin (LMWH) within 12 hours of randomization
* Intravenous low dose thrombolysis (20 mg of rtPA, Alteplase) over 6 hours plus UFH or low molecular weight heparin (LMWH).
* UFH or low molecular weight heparin (LMWH) only (with option for conventional thrombolysis according to local protocols for hemodynamic deterioration) Design: Regional collaborative, randomized trial with 1:1:1 allocation of 210 patients with acute intermediate-high risk PE with no absolute contraindications to thrombolysis

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Informed consent for trial participation
3. Intermediate high-risk PE according to ESC criteria
4. Thrombus visible in main, lobar or segmental pulmonary arteries on CT angiography
5. 14 days of symptoms or less

Exclusion Criteria:

1. Altered mental state (GCS < 14)
2. No qualifying CT angiography performed (> 24 hour since CT angiography)
3. Females of child bearing potential, unless negative HCG test is present
4. Thrombolysis for PE within 14 days of randomization
5. Thrombus passing through patent Foramen Ovale (risk of paradoxical embolism)
6. Ongoing oral anticoagulation therapy (heparins, aspirin, antiplatelet therapy and NOAC allowed)
7. Comorbidity making 6 months survival unlikely
8. Absolute contraindications for thrombolysis

   1. Hemorrhagic stroke or stroke of unknown origin at any time
   2. Ischemic stroke in the preceding 6 months
   3. Central nervous system damage or neoplasms
   4. Recent major trauma/surgery/head injury in the preceding 3 weeks
   5. Gastrointestinal bleeding within the last month
   6. Known bleeding risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Miller score comparing low dose thrombolysis and heparin alone groups | at 48 to 96 hours post randomization
  Reduction in Miller Score and on follow-up (48-96 h) CT pulmonary Angiography comparing low-dose rtPA (±USAT) to UFH/LMWH group (p<0.01, N=210)
Reduction i Miller score comparing low dose thrombolysis by iv and by USATgroups | at 48 to 96 hours post randomization
  reduction in Miller Score and on follow-up (48-96 h) CT pulmonary Angiography comparing low-dose rtPA by USAT to iv, p<0.04, N=140)

SECONDARY OUTCOMES:
Incidence of bleeding complications | Until hospital discharge, on average 1 week
  Bleeding complications (major and minor bleeding complication according the TIMI classification)
Length of stay of index admission | End of study, expected to be 5 years
  Duration of index admission, including hospital based rehabilitation
Dyspnea index by visual analogue scale | End of study, expected to be 5 years
  Dyspnea index (Visual analog scale) after 48-96 h and after 3 months
Change in oxygen supplement (FiO2) | at 48 to 96 hours post randomization
  FiO2 (in %)
Mortality rate | End of study, expected to be 5 years
  Mortality in the three groups (log-rank), and hazard ratio in multivariable analysis using the UFH/LMWH as reference
Incidence of Pulmonary Hypertension | 3 months follow-up
  Incidence of TR gradient > 40 mmHg at 3 months follow-up echocardiography
6 minute walk distance af follow-up | 3 months follow-up
  6 minute walk distance at 3 months follow-up visit
Health related Quality of Life (PEmb-QoL) | 3 months follow-up
  Health related Quality of Life at 3 months follow-up using PEmb-QoL (Pulmonary Embolism Quality of Life) ranging from 0 to 100, higher score indicating worse Quality of Life
Health related Quality of Life (EQ-5D-5L) | 3 months follow-up
  5Q-5D-5L (EuroQoL 5 dimension, 5 level questionnaire, ranging from -0.59 to 1, where 1 is the best possible health state)

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital Gentofte, Gentofte Municipality, Capital Region
  - Copenhagen University Hospital Bispebjerg Hospital, Bispebjerg
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Copenhagen University Hospital, Herlev Gentofte Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Undecided
Main trial database

REFERENCES:
- [Derived] Kjaergaard J, Bang LE, Sonne-Holm E, Wiberg S, Holmvang L, Lassen JF, Sorensen R, Hofsten DE, Ulriksen PS, Jawad S, Palm P, Soe C, Ersboll MK, Boesgaard S, Moller JE, Thune JJ, Hassager C, Tilsted HH, Lonborg J, Egstrup M, Kristiansen OP, Seven E, Lindholm MG, Eskesen K, Fano S, Carlsen J. Randomized trial of low-dose -, ultrasound assisted thrombolysis or heparin for pulmonary embolism. Cardiovasc Res. 2026 Jan 29:cvag038. doi: 10.1093/cvr/cvag038. Online ahead of print. PMID 41610160
- [Derived] Kjaergaard J, Carlsen J, Sonne-Holm E, Wiberg S, Holmvang L, Lassen JF, Sorensen R, Hofsten D, Ulriksen PS, Jawad S, Palm P, Thune JJ, Hassager C, Kristiansen OP, Eskesen K, Fano S, Bang LE. A randomized trial of low-dose thrombolysis, ultrasound-assisted thrombolysis, or heparin for intermediate-high risk pulmonary embolism-the STRATIFY trial: design and statistical analysis plan. Trials. 2024 Dec 28;25(1):853. doi: 10.1186/s13063-024-08688-4. PMID 39732696